CLINICAL TRIAL: NCT02863003
Title: Multicenter Database of Patients With Germ Cell Tumor in Order to Characterize Clinicopathologically and to Evaluate Cancer Treatment Outcomes
Brief Title: Multicenter Database of Patients With Germ Cell Tumor
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: LACOG 0515
Record Dates: First submitted 2016-07-07; First posted 2016-08-11 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-08

CONDITIONS: Neoplasms, Germ Cell and Embryonal
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 16 Years

SUMMARY:
Retrospective and prospective cohort of patients with germ cell tumor in treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to create a multicenter database in order to characterize epidemiologically and clinicopathologically patients with germ cell tumor and evaluate the prognosis and clinical outcomes during cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with diagnosis of testicular, retroperitoneum or mediastinal primary tumor.
* Histological confirmation of germ cell tumor or clinical condition based on the elevation of tumor markers (AFP, HCG e/ou DHL) associated to testicular mass or/and retroperitoneal lymphnode enlargement or/and mediastinal mass.
* Medical records of the disease and treatment

Exclusion Criteria:

* Female patients diagnosed with ovary germ cell tumor
* Male patients diagnosed with germ cell tumor in other locations.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with diagnosis of testicular, retroperitonium or mediastinal primary tumor.
Sampling Method: Non-Probability Sample
Enrollment: 1315 (Actual)
Dates: Start 2016-09; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Brazilian multicenter database in order to collect and analyze data from diagnosis and treatment of patients with germ cell tumor | From 2000 to 2025

SECONDARY OUTCOMES:
Description of demographic characteristics of testicular germ cell tumor patients in Brazil | From 2000 to 2025
The clinical and pathological characteristics of testicular germ cell tumor patients in Brazil. | From 2000 to 2025
Treatment according to staging and relapse of patients diagnosed with testicular germ cell tumor in Brazil | From 2000 to 2025
Disease free survival of patients diagnosed with germ cell tumor stage 1. | From 2000 to 2025
Overall survival of patients diagnosed with germ cell tumor stage 1. | From 2000 to 2025
Disease free survival of patients diagnosed with germ cell tumor stages 2 and 3. | From 2000 to 2025
Overall survival of patients diagnosed with germ cell tumor stages 2 and 3. | From 2000 to 2025
International prognostic factors in patients with advanced germ cell tumor (stages 2 and 3) stablished by the International Germ Cell Cancer Collaborative Group in brazilian patients. | From 2000 to 2025
Treatment outcome in different populations: in patients with brain metastasis, patients with germinative tumor extragonodal, surgery outcome in patients with nonseminomous tumor and ressection of residual lesion after chemotherapy | From 2000 to 2025
Disease free survival of patients diagnosed with disease relapse after first line chemotherapy | From 2000 to 2025
Overall survival of patients diagnosed with disease relapse after first line chemotherapy | From 2000 to 2025
Prognostic model after first line treatment failure with cisplatin, stablished by the International Prognostic Factors Study Group in brazilian patients. | From 2000 to 2025

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Werutsky, MD, Study Director — Latin American Cooperative Oncology Group; Diogo Bastos, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (4):
- Brazil (4):
  - CPO - Pucrs, Porto Alegre, Rio Grande do Sul
  - Hospital Israelita Albert Einstein, São Paulo
  - Hospital São José, São Paulo
  - ICESP, São Paulo